CLINICAL TRIAL: NCT04688762
Title: The E-consult Application for Patients With Breast Cancer: Interest in Empathy and Empowerment of Patients.
Acronym: e-CONSULT
Status: Completed | Type: Observational
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A02045-34
Record Dates: First submitted 2020-12-24; First posted 2020-12-30 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer; Surgery
Keywords: empathy
MeSH Terms: conditions — Breast Neoplasms | interventions — Equipment and Supplies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group without the e-consult tool: standard consultation
- Group with the e-consult tool: The e-consult tool is a digital application developed and designed by the Center François Baclesse, This tool is a consultation support to explain the surgical management of the patient.
  Interventions: Other: e-consult application (tool)

INTERVENTIONS:
Other: e-consult application (tool) — A numeric application used as a support in consultation to explain the surgical management of the patient.
  Groups: Group with the e-consult tool

SUMMARY:
Demonstrate that the use of this application in consultation could improve the empathy perceived of the doctors by the patients after the consultation.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years old
* Patient referred for first consultation for surgery
* Patient referred for a breast tumorectomy and axillary sentinel node
* No patient opposition to participating in this study

Exclusion Criteria:

* Non-surgical management
* Management by any surgery other than breast tumorectomy and axillary sentinel node
* Any associated medical, social or psychopathological condition that could compromise the patient's ability to participate in the study
* Patient deprived of liberty or under guardianship
* Person subject to legal protection or unable to express their consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with breast cancer with surgery indication
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2020-12-24 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
Demonstrate that the use of this application in consultation could improve the empathy perceived of the doctors by the patients after the consultation. | before surgery
  The average obtained in the CARE questionnaire by patients (score [10-50])

CONTACTS AND LOCATIONS:
Locations (1):
- Centre François Baclesse, Caen, France

IPD SHARING:
Plan to Share IPD: No